CLINICAL TRIAL: NCT06047951
Title: Brain Low-risk Aneurysm Stereotactic Radiosurgical Trial: A Phase 2 Nonrandomized Controlled Trial
Brief Title: Brain Low-risk Aneurysm Stereotactic Radiosurgical Trial
Acronym: BLAST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr David Mathieu (Other)
Collaborators: Université de Sherbrooke (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor-Investigator, Dr David Mathieu, Director of the Division of Neurosurgery, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Organization: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4097
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Intracranial Aneurysm
Keywords: brain aneurysm, radiosurgery, intracranial aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: The study population will consist of adult men and women with a CTA-proven UIA under 7 mm who were advised to not undergo treatment because of its low rupture risk. The sample will consist of consecutively enrolled patients seen for a vascular neurosurgical consult or follow-up in the outpatient clinic of participating centers. All eligible patients will be offered to participate in the study at the next follow-up. Enrolled patients will then decide if they want to undergo SRS or if they prefer to continue being managed expectantly. Patients who decide to undergo SRS will be treated with radiosurgery according to the study protocol, while patients who decline SRS will be enrolled in a control, prospective, observational cohort with the same follow-up protocol as the SRS cohort. Furthermore, patients harbouring multiple UIAs will only be treated for one lesion. There will be no randomization or blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SRS group (Experimental): Participants in the SRS group will receive the intervention described earlier, consisting of a Gamma Knife radiosurgery, and undergo the same follow-up exams (radiological and clinical) as participants of the control group.
  Interventions: Procedure: Stereotactic RadioSurgery (SRS)
- Control group (No Intervention): The medical care will consist of observation for any element that may indicate an increased risk of rupture, like aneurysm growth or instability in shape.

INTERVENTIONS:
Procedure: Stereotactic RadioSurgery (SRS) — All treatments will be performed using the Gamma Knife Perfexion or Icon system (Elekta). The following treatment parameters will be used:
  * The head will be immobilized using a stereotactic Leksell Model G frame, installed using local protocols
  * Targeting will be performed by using a stereotactic CTA. No MRI will be performed.
  * Only one aneurysm will be treated per patient
  * The aneurysm, including its neck, will be contoured and targeted using a combination of 4mm isocenters as deemed appropriate by the treating team
  * A prescription dose of 25 Gy at the margin of the target will be used
  * The maximal dose on optic pathways will be kept below 10 Gy
  * The brainstem 12-Gy volume will be kept below 1cc
  Other Names: Gamma Knife SRS
  Arms: SRS group

SUMMARY:
The goal of this clinical trial is to confirm the feasibility and safety of performing radiosurgery on unruptured, low-risk aneurysms in humans.

Participants will choose if they want to undergo radiosurgery or not. Participants who choose not to have radiosurgery will be assigned to the observational group. Participants who choose to have radiosurgery performed will be assigned to the radiosurgery group. Participants in both groups will attend an initial exam session as well as four follow-up sessions:

Day 0

* Initial questionnaire
* CTA scan
* MRI
* Radiosurgery performed on patients in the radiosurgery group

  6 months
* CTA scan
* Follow-up questionnaire

  12 months
* CTA scan
* MRI
* Follow-up questionnaire

  24 months
* CTA scan
* Follow-up questionnaire

  36 months
* CTA scan
* MRI
* Follow-up questionnaire

Researchers will compare the observational group and the radiosurgery group to see if there is a difference in the incidence of aneurysm rupture during the study period (3 years). The hypothesis is that radiosurgery should not increase the risk of aneurysm rupture.

DETAILED DESCRIPTION:
This study is designed as a phase 2, two-arm, open label trial comparing a group undergoing stereotactic radiosurgery (SRS) to a control, observational group.

Sample size

This is a phase 2 safety and feasibility study, therefore, powering for effectiveness is not required. The initial target sample size is 20 patients in the SRS group and 20 patients in the control group. This should be sufficient to detect complications associated with SRS that exceed a 5% incidence rate and assess if obliteration can be achieved in some patients.

If the goal of 20 patients is reached in one of the groups, the investigatrors will recruit only in the second group, until the goal of 20 patients per group is reached.

Setting and screening

Potentially eligible patients will be screened by vascular neurosurgeons at the time of neurosurgical consult or follow-up in the outpatient clinic. The physician will inform the patient of the existence of the research project and offer him to meet the research nurse. If the patient agrees, the nurse will meet the patient within two hours of the consult. The research nurse will present the study, confirm his eligibility and obtain written consent. A copy of the consent form will be given to the patient and another will be stored in the patients' research chart. The subject is free to terminate his participation in the study at any time.

Variables and data collection

The measured variables are presented below.

- Treatment (Binary: SRS/None, Independent variable)

Demographic and baseline variables data

* Age at enrollment (Continuous (years), Initial questionnaire)
* Gender (Binary: Female/Male, Initial questionnaire)
* Diabetes mellitus (Binary: No/Yes, Initial questionnaire)
* Hypertension (Binary: No, Yes, Initial questionnaire)
* Active smoking (Binary: No/Yes, Initial questionnaire, To be considered inactive, the subject must have stopped smoking for more than 4 weeks.)
* Cumulative smoking (Continuous: pack-year, Initial questionnaire)
* Current alcohol use (Continuous: number of alcoholic beverages per week, Initial questionnaire)
* Any pertinent factor (Free text, Initial questionnaire)

Clinical presentation

- How was the aneurysm discovered? (Categorical: Incidental discovery/Screening imaging because of family history/Other (please specify), Initial questionnaire)

CTA scan at enrolment

* Date of the CTA scan (Date, Medical record)
* Aneurysm location (Categorical: A1/ACom/A2/M1/MCA bifurcation/M2/Anterior choroidal/Ophthalmic/Superior hypophysial/PCom, CTA scan at enrolment)
* Side of aneurysm (Categorical: Right/Left/Midline, CTA scan at enrolment)
* Aneurysm volume (Continuous (mm3), CTA scan at enrolment, Volume will be measured by segmentation)
* Aneurysm height (z) (Continuous (mm), CTA scan at enrolment, Measured in the longest axis, perpendicular to the neck)
* Aneurysm width (x) (Continuous (mm), CTA scan at enrolment, Measured in the longest axis, perpendicular to the height)
* Aneurysm width (y) (Continuous (mm), CTA scan at enrolment, Measured in the longest axis, perpendicular to both height and width (x))
* Aneurysm neck diameter (Continuous (mm), CTA scan at enrolment)
* Aneurysm surface area (Continuous (mm2), CTA scan at enrolment, Computed from the segmented volume)
* Aneurysm aspect ratio (AR) (Continuous, AR is a 2D shape indicator that is a good predictor of rupture risk22)
* Aneurysm non-sphericity index (NSI) (Continuous, NSI is currently the best predictor of rupture amongst shape indices. It is a 3D indicator of how much deviation in shape there is between the aneurysm and a sphere of equal volume)

SRS treatment

* Treatment date (Date, Medical record)
* Was treatment completely administered? (Binary: Yes/No, Medical record)
* Total treatment time (Continuous (min), GammaPlan record)
* Beam-on time (Continuous (min), GammaPlan record)
* Maximum dose (Continuous (Gy), GammaPlan record)
* Margin dose (Continuous (Gy), GammaPlan record)
* Isodose line (Continuous (%), GammaPlan record)
* Nb of isocenters (Continuous, GammaPlan record)
* Treatment volume (Continuous (mm3), GammaPlan record)
* Brainstem 12 Gy volume (Continuous (mm3), GammaPlan record)
* Maximum optic chiasm dose (Continuous (Gy), GammaPlan record)

Radiological follow-up (CTA at 6, 12, 24 and 36 months after SRS, MRI at 12 and 36 months after SRS)

* Date of follow-up (Date, CTA)
* Complete aneurysm obliteration? (Binary: Yes/No, CTA)
* Aneurysm rupture? (Binary: Yes/No, CTA, If aneurysm rupture occurs, an aneurysm rupture report must be completed)
* Aneurysm volume (Continuous (mm3), CTA, Volume will be measured by segmentation)
* Aneurysm height (z) (Continuous (mm), CTA, Measured in the longest axis, perpendicular to the neck)
* Aneurysm width (x) (Continuous (mm), CTA, Measured in the longest axis, perpendicular to the height)
* Aneurysm width (y) (Continuous (mm), CTA, Measured in the longest axis, perpendicular to both height and width (x))
* Aneurysm neck diameter (Continuous (mm), CTA)
* Aneurysm surface area (Continuous (mm2), CTA, Computed from the segmented volume.)
* Aneurysm aspect ratio (AR) (Continuous, AR is a 2D shape indicator that is a good predictor of rupture risk22)
* Aneurysm non-sphericity index (NSI) (Continuous, NSI is currently the best predictor of rupture amongst shape indices. It is a 3D indicator of how much deviation in shape there is between the aneurysm and a sphere of equal volume.)
* Evidence of adverse radiation-induced effect? (Binary: Yes (please detail)/No, MRI)

Clinical follow-up at 6, 12, 24 and 36 months

* Date of the clinical follow-up (Date, Medical record)
* Aneurysm rupture (Binary: Yes/No, Medical record)

If the aneurysm did rupture:

* Date of rupture (Date, Medical record)
* SAH grade (Categorical: I/II/III/IV/V, Medical record, As defined by the World Federation of Neurosurgical Societies (WFNS))
* Treatment complications:
* New neurological deficit (Categorical: None/Grade 1/Grade 2/Grade 3, Medical record and follow-up questionnaire, As graded by CTCAE v5)
* Cerebral edema (Categorical: None/Grade 3/Grade 4/Grade 5, Medical record and follow-up questionnaire, As graded by CTCAE v5)
* Stroke (Categorical: None/Grade 1/Grade 2/Grade 3/Grade 4/Grade 5, Medical record and follow-up questionnaire, As graded by CTCAE v5)
* Radiation necrosis (Categorical: None/Grade 1/Grade 2/Grade 3/Grade 4/Grade 5, Medical record and follow-up questionnaire, As graded by CTCAE v5)
* De novo seizure (Categorical: None/Grade 1/Grade 2/Grade 3/Grade 4/Grade 5, Medical record and follow-up questionnaire, As graded by CTCAE v5)
* Increase in seizure frequency (Binary: Yes/No, Medical record and follow-up questionnaire)
* Headache (Categorical: None/Grade 1/Grade 2/Grade 3, Medical record and follow-up questionnaire, As graded by CTCAE v5)
* Facial pain Categorical: None/Grade 1/Grade 2/Grade 3, Medical record and follow-up questionnaire, As graded by CTCAE v5)
* Other (specify) (Categorical: None/Grade 1/Grade 2/Grade 3/Grade 4/Grade 5, Medical record and follow-up questionnaire, As graded by CTCAE v5)

If so:

* Date of first symptoms (Date, Medical record and follow-up questionnaire)
* Description of the complication (Free text, Medical record and follow-up questionnaire)
* Treatment (Categorical: Successfully treated/Treated, but symptoms persist/Not treated, but symptoms subsided/Not treated and symptoms persist, Medical record and follow-up questionnaire)
* Description of the treatment (Free text, Medical record)
* Date of last symptoms (if symptoms subsided) (Date, Medical record and follow-up questionnaire)

Other treatments after SRS:

- Surgical intervention (Binary: Yes/No, Medical record)

If yes:

* Date of surgery (Date, Medical record)
* Surgical urgency (Categorical: Elective surgery/Urgent surgery, Medical record, An urgent surgery is a procedure that could not wait until the next day.)
* Surgery details (Medical record)
* Endovascular procedure (Binary: Yes/No, Medical record)

If yes:

* Date of procedure (Date, Medical record)
* Urgency of procedure (Categorical: Elective surgery/Urgent surgery, Medical record, An urgent endovascular surgery is a procedure that could not wait until the next day.)
* Procedure details (Medical record)

Death (Binary: Yes/No, Medical record)

If yes:

- Date of death (Date, Medical record)

Measurement instruments

CTA scan

CTA scanning is commonly used in clinical practice for the diagnosis and follow-up of intracranial aneurysms because of its non-invasive nature8. It is an X-Ray imaging technique allowing tridimensional reconstruction of the skull and its content, with reported sensitivities ranging from 0.77 to 0.97 and specificities ranging from 0.87 to 1.00 for intracranial aneurysms12. The test requires the patient to go to the department of radiology where the scanner is located. The scan itself takes between 15-30 minutes during which the patient is lying on his back. The test is not painful, but some claustrophobic patients might feel temporarily anxious while inside the scanner.

CTA scans in the protocol require intravenous injections of iodine solution to make blood vessels opaque. This step requires the installation of an IV line for the duration of the scan. If the patient is allergic to the iodine solution, a desensitization protocol will be initiated with antihistamines and corticosteroids. In case of renal failure (eGFR < 60mL/min), patients need to be hyperhydrated or another modality considered (MRA or DSA).

Following the scan, the subject can return to his home.

The study's radiological follow-up schedule has been conceived to follow the standard radiological follow-up performed for UIAs at the CHUS. Therefore, while the follow-up CTA scans will be prescribed by the research nurse to comply with the study's standardized schedule, there will be no additional test required relative to a patient observed at the CHUS outside of this trial.

Aneurysm volume and dimensions will be measured using segmentation facilities within the Osirix 6.5 (Pixmeo, Genève, Suisse) software. Radiological obliteration will be defined as the absence of a residual, measurable arterial wall dilation where the aneurysm used to be. Once the study is completed, official measurements used for the analysis of the primary and secondary outcomes will be performed by a single, independent and blinded radiologist.

Magnetic Resonance Imaging (MRI)

MRI uses a strong magnetic field, proton density and radiofrequency waves to generate detailed anatomical images non-invasively. Because of its superior image definition, it is the preferred method to assess brain parenchyma integrity. Patients are asked to lie in a tube-shaped magnet and hold still for 20-30 min. The test is not painful, but some claustrophobic patients may feel temporarily anxious while inside the scanner.

MRI sequences used in this protocol include a standard T1 weighted sequence with and without contrast enhancement, a FLAIR sequence and a diffusion weighted sequence. Thus, installation of an IV line for the duration of the scan and administration of gadolinium to enhance the visibility of certain structures is required. If the patient is allergic to the gadolinium solution, a desensitization protocol will be initiated with antihistamines and corticosteroids. In case of severe renal failure (eGFR < 30 mL/min), patients will need to be hyperhydrated or images will be taken without the administration of contrast agent.

Patients may resume their activities immediately after the scan.

The study's radiological follow-up schedule has been conceived to follow the standard radiological follow-up performed for UIAs at the CHUS. Therefore, while the follow-up MRI will be prescribed by the research nurse to comply with the study's standardized schedule, there will be no additional test required relative to a patient observed at the CHUS outside of this trial.

Study flow

Identification and enrolment

* Identification of potentially eligible subjects is performed at the time of consult or follow-up by the neurovascular surgeon. Upon patient agreement, the research nurse is called;
* Enrolment is performed by the research nurse who will meet the patient within 2 hours of the initial consult. The nurse will present the project and obtain written consent. A paper copy of the consent form is given to the patient and another is signed and kept in the patient's research record.

Initial data collection

Following informed consent, the research nurse:

* Completes the initial questionnaire);
* Schedules, under the local PI, the SRS procedure for patients in the SRS group;
* Prescribes, under the local PI, the follow-up CTA scan at 6 months for the control group;

SRS treatment

* SRS is performed on patients in the SRS group.
* The research nurse prescribes, under the local PI, the follow-up CTA scan at 6 months for the SRS group.

Follow-up

At 6 months:

A control CTA scan is performed.

* The research nurse contacts the local PI who will assess aneurysm resolution.
* The research nurse prescribes a control CTA scan and MRI at 12 months.

At 12 months:

* A control CTA scan and MRI are performed
* The research nurse contacts the local PI who will assess aneurysm resolution.
* The research nurse prescribes a control CTA scan at 24 months.

At 24 months:

* A control CTA scan is performed
* The research nurse contacts the local PI who will assess aneurysm resolution.
* The research nurse prescribes a control CTA scan and MRI at 36 months.

At 36 months:

* A control CTA scan and MRI are performed
* The research nurse contacts the local PI who will assess aneurysm resolution.
* The follow-up schedule will be determined at the discretion of the treating physician

Details relative to the conduct of the study

Adverse event monitoring

Adverse events (AE) potentially related to SRS will systematically be documented at each planned follow-up through radiological investigations and follow-up questionnaires.

In addition, treating teams must notify the local PI of any AE potentially linked to SRS within 24 hours of detection. The local PI will inform the coordinating center within 5 days.

A serious AE is an AE with one of the following features:

* Leads to death of the subject;
* Life-threatening for the subject;
* Requires hospital admission or prolongs hospital admission;
* Leads to permanent or significant disability;
* Leads to a permanent, significant or congenital abnormality.

An unexpected event is a complication resulting from SRS that is not mentioned in the treatment's list of complications and side-effects.

There will be a mechanism in place so that research teams will be notified if one of their subjects is admitted so that serious AE can be proactively identified.

Data collection

All data collected as part of this study will be stored in one of the following systems:

Patient's paper research record :

* This is a paper file stored in a locked office by the research nurse within the research center;
* Documents stored in this file include all paper forms, such as: signed consent form, initial questionnaire, any follow-up questionnaires, AE report or aneurysm rupture report
* Patient's hospital medical record: This is the standard medical record of the patient. It will contain all imaging studies performed.

All the collected data will be kept for 25 years following publication of the study results.

Data analysis

Once the last follow-up of the last subject will be performed, data will be compiled onto an excel spreadsheet to perform the pre-planned statistical analyses using SPSS. Data will be analyzed using the statistical tests presented below.

The detailed statistical analysis and computer program will be published before the end of subject enrollment.

Comparison of study characteristics between both groups (SRS vs. control)

* Number of enrolled subjects (Binary, Chi2, Fisher exact test)
* Number of subjects lost in follow-up (Binary, Chi2, Fisher exact test)

Comparison of baseline characteristics between both groups (SRS vs. control)

* Mean age at enrollment (years) (Continuous, Standard deviation, Student T test vs Mann-Withney)
* Gender (% male) (Continuous, Student T test vs Mann-Withney)
* Active smoker (%) (Continuous, Student T test vs Mann-Withney)
* Mean cumulative smoking (pack-years) (Continuous, Standard deviation, Student T test vs Mann-Withney)
* Current alcohol consumption (number of alcoholic beverages per week) (Continuous, Standard deviation, Student T test vs Mann-Withney)
* Mean aneurysm volume at diagnosis (mL) (Continuous, Standard deviation, Student T test vs Mann-Withney)

Effect of the intervention (SRS vs. control group)

* Primary outcome (Continuous, Student T test vs Mann-Withney)
* Aneurysm volume evolution (Series of continuous values, Repeated-measures ANOVA)
* Aneurysm resolution (Binary, Chi2, Fisher exact test)

Risk factors for meeting the primary outcome (primary outcome met vs. not met) for all subjects

Risk factors to be assessed:

* Administered treatment (SRS vs nothing)
* Age
* Current alcohol consumption
* Active smoking
* Hypertension
* Cumulative smoking
* Aneurysm location
* Aneurysm initial volume
* Aneurysm AR
* Aneurysm NSI (Logistic regression)

Risk factors for meeting the primary outcome (primary outcome met vs. not met) for patients in SRS group only

Risk factors to be assessed:

* Treatment volume
* Maximum dose
* Dose rate
* BED (Logistic regression)

Risk factors for aneurysm occlusion at 3 years confirmed by CT-angiography (CTA) for patients in SRS group only

Risk factors to be assessed:

* Age
* Current alcohol consumption
* Active smoking
* Hypertension
* Cumulative smoking
* Aneurysm location
* Aneurysm initial volume
* Treatment volume
* Maximum dose
* Dose rate
* BED (Logistic regression)

Risk factors for endovascular or surgical aneurysm treatment during the latency period for all subjects

Risk factors to be assessed:

* Administered treatment (SRS vs nothing)
* Age
* Current alcohol consumption
* Active smoking
* Hypertension
* Cumulative smoking
* Aneurysm location
* Aneurysm initial volume
* Aneurysm AR
* Aneurysm NSI (Logistic regression)

Risk factors for change in aneurysm volume relative to baseline for patients in SRS group only

Risk factors to be assessed:

* Age
* Current alcohol consumption
* Active smoking
* Hypertension
* Cumulative smoking
* Aneurysm location
* Aneurysm initial volume
* Treatment volume
* Maximum dose
* Dose rate
* BED (Logistic regression)

Risk factors for change in aneurysm shape indices relative to baseline for patients in SRS group only

Risk factors to be assessed:

* Age
* Current alcohol consumption
* Active smoking
* Hypertension
* Cumulative smoking
* Aneurysm location
* Aneurysm initial volume
* Treatment volume
* Maximum dose
* Dose rate
* BED (Logistic regression)

Risk factors for occurrence of any radiation-induced complications for patients in SRS group only

Risk factors to be assessed:

* Age
* Diabetes mellitus
* Current alcohol consumption
* Active smoking
* Cumulative smoking
* Aneurysm location
* Aneurysm initial volume
* Treatment volume
* Maximum dose
* Dose rate
* Margin dose
* BED (Logistic regression)

Safety analysis (SRS vs. control group)

- Stroke (Binary, Chi2, Fisher exact test)

Ethical considerations

Free and informed consent

Consent will be free and informed. Specifically:

* Enrollment will be performed by a research nurse independent from the treating team.
* No pressure will be put on the patient to increase enrollment in the SRS group. This is supported by the fact that there is an equal need for patients in the observational cohort, as there is a need for patients in the interventional group.
* Patients who are unable to consent to their care will not participate in the study.
* The subject can stop the study at any time.
* Participation in the study does not change patient management or access to tests or facilities required for the optimal treatment of his condition.

Risks related to study participation

Some of the risks subjects face are related to their medical condition (UIA) and exist regardless of their participation in the study. These risks include risks related to CTA and MRI scanning and the surgical/endovascular procedures that could be performed. These risks are not discussed in the consent form, because they are not related to study participation.

The risks related to study participation are:

Risks related to SRS treatment (for subjects in the intervention group). This treatment option is well known, already widely used by neurosurgeons and well tolerated. Reported side effects include:

* Headache
* Seizures
* Nausea
* Cerebral oedema
* Focal neurological deficits (depending on treated lesion location)
* Radiation necrosis

The risks related to CTA and MRI scanning are not related to study participation and are not discussed.

Disadvantages related to study participation

Subjects will need to meet with the research nurse on the day of enrollment and patients electing to undergo SRS will need to dedicate a complete day to the procedure.

Confidentiality

Confidentiality will be strictly respected throughout the study. The use of paper charts will limit the potential for a breach in data security, and only denominated data will be transferred in Excel at the time of analysis.

Participant compensation

There is no compensation for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Medical imaging (CTA, MRA or digital substraction angiography) reveals the existence of an asymptomatic unruptured saccular anterior circulation intracranial aneurysm under 7 mm
* Advised by a vascular neurosurgeon to observe rather than undergo endovascular or microsurgical management

Exclusion Criteria:

* Prior history of aneurysmal rupture
* Presence of symptoms that could be attributed to the aneurysm (severe headache, third cranial nerve deficits, or others)
* Imaging features deemed to increase rupture risk as evaluated by the treating physician
* Posterior circulation aneurysm
* Fusiform aneurysm
* Dissecting aneurysm
* Mycotic aneurysm
* Direct contact between the aneurysm and the optic pathways on medical imaging
* Prior coils or clips in the targeted aneurysm or any other aneurysm
* Patient unable to consent
* Patient unable or unlikely to comply with the follow-up schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Between group difference in the incidence of aneurysm rupture during the study period | 3 years from SRS
  The hypothesis is that SRS should not increase this risk.

SECONDARY OUTCOMES:
Incidence of any radiation-induced complications | 3 years
  ex: brain edema, radiation necrosis
Incidence of endovascular or surgical aneurysm treatment during the latency period | 3 years
  Number of patients undergoing treatment
Change in aneurysm volume relative to baseline | 3 years
  Aneurysm volume in cubic millimeters (mm3) and dimensions in millimeters (mm) will be measured using segmentation facilities within the Osirix 6.5 software.
Change in aneurysm shape indices relative to baseline | 3 years
  ex. Nonsphericity index, Aspect ratio, etc.
Aneurysm occlusion confirmed by CT-angiography (CTA) | at 3 years from SRS
  Complete, partial or no occlusion

CONTACTS AND LOCATIONS:
Overall Officials: David Mathieu, MD FRCS(C), Principal Investigator — Service de neurochirurgie, Département de chirurgie, Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers.

REFERENCES:
- [Background] Kleinloog R, de Mul N, Verweij BH, Post JA, Rinkel GJE, Ruigrok YM. Risk Factors for Intracranial Aneurysm Rupture: A Systematic Review. Neurosurgery. 2018 Apr 1;82(4):431-440. doi: 10.1093/neuros/nyx238. PMID 28498930
- [Background] Bonneville F, Sourour N, Biondi A. Intracranial aneurysms: an overview. Neuroimaging Clin N Am. 2006 Aug;16(3):371-82, vii. doi: 10.1016/j.nic.2006.05.001. PMID 16935705
- [Background] Meadowcroft MD, Cooper TK, Rupprecht S, Wright TC, Neely EE, Ferenci M, Kang W, Yang QX, Harbaugh RE, Connor JR, McInerney J. Gamma Knife radiosurgery of saccular aneurysms in a rabbit model. J Neurosurg. 2018 Dec 1;129(6):1530-1540. doi: 10.3171/2017.6.JNS17722. Epub 2018 Jan 12. PMID 29328001
- [Background] Erratum: Management of unruptured intracranial aneurysms. Neurol Clin Pract. 2014 Apr;4(2):98. doi: 10.1212/CPJ.0000000000000019. PMID 29443238
- [Background] Flemming KD, Lanzino G. Management of Unruptured Intracranial Aneurysms and Cerebrovascular Malformations. Continuum (Minneap Minn). 2017 Feb;23(1, Cerebrovascular Disease):181-210. doi: 10.1212/CON.0000000000000418. PMID 28157750
- [Background] Schievink WI. Intracranial aneurysms. N Engl J Med. 1997 Jan 2;336(1):28-40. doi: 10.1056/NEJM199701023360106. No abstract available. PMID 8970938
- [Background] Fusco MR, Ogilvy CS. Surgical and endovascular management of cerebral aneurysms. Int Anesthesiol Clin. 2015 Winter;53(1):146-65. doi: 10.1097/AIA.0000000000000038. No abstract available. PMID 25551747
- [Background] Brown RD Jr, Broderick JP. Unruptured intracranial aneurysms: epidemiology, natural history, management options, and familial screening. Lancet Neurol. 2014 Apr;13(4):393-404. doi: 10.1016/S1474-4422(14)70015-8. PMID 24646873
- [Background] Burns JD, Brown RD Jr. Treatment of unruptured intracranial aneurysms: surgery, coiling, or nothing? Curr Neurol Neurosci Rep. 2009 Jan;9(1):6-12. doi: 10.1007/s11910-009-0002-0. PMID 19080747
- [Background] Truelsen T, Bonita R, Duncan J, Anderson NE, Mee E. Changes in subarachnoid hemorrhage mortality, incidence, and case fatality in New Zealand between 1981-1983 and 1991-1993. Stroke. 1998 Nov;29(11):2298-303. doi: 10.1161/01.str.29.11.2298. PMID 9804637
- [Background] Qureshi AI, Suri MF, Nasar A, Kirmani JF, Divani AA, He W, Hopkins LN. Trends in hospitalization and mortality for subarachnoid hemorrhage and unruptured aneurysms in the United States. Neurosurgery. 2005 Jul;57(1):1-8; discussion 1-8. doi: 10.1227/01.neu.0000163081.55025.cd. PMID 15987534
- [Background] Brisman JL, Song JK, Newell DW. Cerebral aneurysms. N Engl J Med. 2006 Aug 31;355(9):928-39. doi: 10.1056/NEJMra052760. No abstract available. PMID 16943405
- [Background] Molyneux AJ, Kerr RS, Yu LM, Clarke M, Sneade M, Yarnold JA, Sandercock P; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group. International subarachnoid aneurysm trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomised comparison of effects on survival, dependency, seizures, rebleeding, subgroups, and aneurysm occlusion. Lancet. 2005 Sep 3-9;366(9488):809-17. doi: 10.1016/S0140-6736(05)67214-5. PMID 16139655
- [Background] Wiebers DO, Whisnant JP, Huston J 3rd, Meissner I, Brown RD Jr, Piepgras DG, Forbes GS, Thielen K, Nichols D, O'Fallon WM, Peacock J, Jaeger L, Kassell NF, Kongable-Beckman GL, Torner JC; International Study of Unruptured Intracranial Aneurysms Investigators. Unruptured intracranial aneurysms: natural history, clinical outcome, and risks of surgical and endovascular treatment. Lancet. 2003 Jul 12;362(9378):103-10. doi: 10.1016/s0140-6736(03)13860-3. PMID 12867109
- [Background] Froelich JJ, Neilson S, Peters-Wilke J, Dubey A, Thani N, Erasmus A, Carr MW, Hunn AW. Size and Location of Ruptured Intracranial Aneurysms: A 5-Year Clinical Survey. World Neurosurg. 2016 Jul;91:260-5. doi: 10.1016/j.wneu.2016.04.044. Epub 2016 Apr 20. PMID 27108026
- [Background] Starke RM, Kano H, Ding D, Lee JY, Mathieu D, Whitesell J, Pierce JT, Huang PP, Kondziolka D, Yen CP, Feliciano C, Rodgriguez-Mercado R, Almodovar L, Pieper DR, Grills IS, Silva D, Abbassy M, Missios S, Barnett GH, Lunsford LD, Sheehan JP. Stereotactic radiosurgery for cerebral arteriovenous malformations: evaluation of long-term outcomes in a multicenter cohort. J Neurosurg. 2017 Jan;126(1):36-44. doi: 10.3171/2015.9.JNS151311. Epub 2016 Mar 4. PMID 26943847
- [Background] Kim BS, Kim KH, Lee MH, Lee JI. Stereotactic Radiosurgery for Brainstem Cavernous Malformations: An Updated Systematic Review and Meta-Analysis. World Neurosurg. 2019 Oct;130:e648-e659. doi: 10.1016/j.wneu.2019.06.183. Epub 2019 Jul 2. PMID 31276856
- [Background] Grady C, Gesteira Benjamin C, Kondziolka D. Radiosurgery for dural arteriovenous malformations. Handb Clin Neurol. 2017;143:125-131. doi: 10.1016/B978-0-444-63640-9.00012-6. PMID 28552134
- [Background] Schneider BF, Eberhard DA, Steiner LE. Histopathology of arteriovenous malformations after gamma knife radiosurgery. J Neurosurg. 1997 Sep;87(3):352-7. doi: 10.3171/jns.1997.87.3.0352. PMID 9285598
- [Background] Lan Z, Li J, You C, Chen J. Successful use of Gamma Knife surgery in a distal lenticulostriate artery aneurysm intervention. Br J Neurosurg. 2012 Feb;26(1):89-90. doi: 10.3109/02688697.2011.591949. Epub 2011 Jul 18. PMID 21767129
- [Background] Liscak R, Vymazal J, Chytka T. Gamma Knife Radiosurgery of Distal Aneurysm: A Case Series. Stereotact Funct Neurosurg. 2021;99(5):381-386. doi: 10.1159/000513956. Epub 2021 Mar 17. PMID 33730736
- [Background] Raghavan ML, Ma B, Harbaugh RE. Quantified aneurysm shape and rupture risk. J Neurosurg. 2005 Feb;102(2):355-62. doi: 10.3171/jns.2005.102.2.0355. PMID 15739566
- [Background] Ding D, Xu Z, Starke RM, Yen CP, Shih HH, Buell TJ, Sheehan JP. Radiosurgery for Cerebral Arteriovenous Malformations with Associated Arterial Aneurysms. World Neurosurg. 2016 Mar;87:77-90. doi: 10.1016/j.wneu.2015.11.080. Epub 2015 Dec 28. PMID 26732956
- [Background] Kim M, Pyo S, Jeong Y, Lee S, Jung Y, Jeong H. Gamma Knife surgery for intracranial aneurysms associated with arteriovenous malformations. J Neurosurg. 2006 Dec;105 Suppl:229-34. doi: 10.3171/sup.2006.105.7.229. PMID 18503361
- [Background] Vymazal J, Liscak R, Novotny J Jr, Janouskova L, Vladyka V. The role of Gamma Knife radiosurgery in arteriovenous malformation with aneurysms. Stereotact Funct Neurosurg. 1999;72 Suppl 1:175-84. doi: 10.1159/000056454. PMID 10681706